CLINICAL TRIAL: NCT07041398
Title: Horizontal Ridge Augmentation Using Sausage Technique: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Berkay Tokuç, Associate Professor, Kocaeli University
Other Study IDs: 2023/384
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Alveolar Bone Grafting; Guided Bone Regeneration; Bone Gain
Keywords: Alveolar bone augmentation; Dental implant; Guided bone regeneration; Horizontal bone gain; Sausage technique

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study investigates the outcomes of the sausage technique, a contemporary modification of guided bone regeneration (GBR), for the augmentation of severely horizontally deficient alveolar ridges (<4 mm width). The technique, originally introduced by Urban and colleagues, uses multiple fixation pins to enhance membrane stability and maintain graft volume through a tension dome effect.

In this study, a total of 23 patients underwent horizontal ridge augmentation using the sausage technique, with bone measurements assessed at 2, 4, and 6 mm apical to the crest using CBCT imaging at preoperative (T0), early postoperative (T1), and late postoperative (T2) stages. The study quantitatively analyzed both horizontal bone gain (T2-T0) and bone resorption (T1-T2) during the healing period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knife-edge alveolar ridges, classified as Class IV according to the Cawood and Howell classification, who underwent ridge augmentation using the sausage technique
* Patients aged 18 or older with fully developed bone
* Patients who had regular clinical and radiographic follow-up after the procedure, with a minimum follow-up period of six months

Exclusion Criteria:

* Patients with systemic conditions (such as osteoporosis, cancer, immunosuppression, hyperparathyroidism, or hyperthyroidism) or a history of medications (including intravenous or oral bisphosphonates, immunosuppressants, or chemotherapy) that could interfere with bone healing
* Patients with a history of radiotherapy to the head or neck region
* Patients classified as ASA III or ASA IV
* Patients who were active smokers at the time of surgery
* Patients whose pre- or postoperative CBCT scans were of low image quality or affected by artefacts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, patient follow-up forms and cone-beam computed tomography (CBCT) scans taken during the pre- and postoperative periods were retrospectively reviewed from the archive of the Department of Oral and Maxillofacial Surgery at Kocaeli University Faculty of Dentistry. All procedures had been performed by the same team (B.T. and Z.D.). Among these records, patients who presented with total or partial edentulism in either jaw and received the sausage technique to treat horizontal alveolar bone deficiency were selected for inclusion.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Amount of horizontal bone gain postoperatively | Within1 week after the collection of patient data
Amount of horizontal bone resorption postoperatively | Within 5 to 7 months postoperatively
Amount of vertical bone resorption postoperatively | Within 5 to 7 months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Faculty of Dentistry, Kocaeli, Başiskele, Turkey (Türkiye)